CLINICAL TRIAL: NCT02143375
Title: Efficacy of810 nm Diode Laser on Gingival Pigmentation
Brief Title: Gingival Depigmentation by Diode Laser
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Somayyeh Babaei, Dr, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mbakhshi
Record Dates: First submitted 2014-04-28; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Laser-induced Hypopigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 810 Diode Laser (Experimental): 810 nm Diode Laser, contact, continuous wave,320micron,
  Interventions: Device: 810 Diode Laser

INTERVENTIONS:
Device: 810 Diode Laser — The 810-nm diode laser has energy and wavelength characteristics that specially target the soft tissues. It has an affinity for hemoglobin and melanin, so it is an excellent soft tissue laser and is applicated for cutting and coagulating gingival tissue.Today,sparse studies have been published assessing physiologic gingival pigmentation using diode laser,therefore the aim of this study was to evaluate the effect of diode laser on the treatment of gingival pigmentation in adult patients.

SUMMARY:
Physiologic gingival pigmentation(PGP) is the most common type of gingival pigmentation and cosmetic concern particularly in gummy smile patients. Laser therapy is an effective and noninvasive treatment option. The aim of this study was to evaluate the efficacy of diod laser on the treatment of PGP in patients.

DETAILED DESCRIPTION:
Preoperative and postoperative photographic and clinical observations about the gingival melanin pigmentation were made according to Dummett-Gupta Oral Pigmentation Index scoring criteria given by Dummett C.O. in 1964 The investigators classified pigmented gingiva in patients as:

1. Mild:Pink to slightly brown
2. Moderate:Deep brown or black
3. Severe:Mixed in color Score in each tooth was taken including one full inter dental papilla. Observations were made in natural light. The assessment of the scoring of the pigmentation index were done by all the three examiners, and the agreed upon score was assigned to prevent individual variations.

The investigators compared the intensity of pigmentation in each patient in recall sessions after 1month and 3mounth postoperative.

ELIGIBILITY:
Inclusion Criteria:

* 19 adult patients who had been referred to oral medicine department of Shahid Beheshti dental school with the chief complaint of melanin pigmentation were selected for inclusion in this study.

Exclusion Criteria:

1. Hyperpigmentation that was associated with systemic disease or drug administration,disease that could compromise wound healing (uncontrolled diabetes, autoimmune disease)
2. Pregnancy or lactation
3. Evidence of relationship between hyperpigmentation and malignancy
4. History of previous treatment of hyperpigmentation
5. Smoking
6. Periodontal problems

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
improvement of gingival pigmentation | 1 month
  standard digital photographs were taken preoperative,1 month after laser therapy.

SECONDARY OUTCOMES:
changes in pigmentation based on standard digital photographs and index of Dummett et al. | 3month
  standard digital photographs were taken 3 months postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Mahin Bakhshi, DDS.MS, Study Chair — Associate Professor of Oral Medicine Department ,Shahid Beheshti Medical University
Locations (1):
- Shahid Beheshti medical university,Dental Faculty, Tehran, Tehran Province, Iran